CLINICAL TRIAL: NCT06139588
Title: Comparative Study of the Efficacy and Risk Profile of Two Animal-derived Acellular Dermal Matrices in Patients Undergoing Mastectomy, Radiotherapy and Implant-based Reconstruction
Brief Title: Comparative Analysis of Two Animal-derived ADMs in Irradiated Implant-based Reconstruction
Acronym: RTADM
Status: Completed | Type: Observational
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: UID4321
Record Dates: First submitted 2023-11-15; First posted 2023-11-18 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-10

CONDITIONS: Breast Implant; Complications; Breast Implant Infection; Implant Capsular Contracture; Breast Seroma; Breast Implant Protrusion; Breast Cancer
Keywords: implant-based; breast reconstruction; adm; radiation therapy; irradiated breast
MeSH Terms: conditions — Implant Capsular Contracture; Breast Neoplasms | interventions — Mammaplasty

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- POST QUART NATIVE: Native adm used in the setting of mastectomy and implant reconstruction after QUART
  Interventions: Device: acellular dermal matrix implant for breast reconstruction
- POST QUART VERITAS: Veritas adm used in the setting of mastectomy and implant reconstruction after QUART
  Interventions: Device: acellular dermal matrix implant for breast reconstruction
- POST EXPANDER NATIVE: Native adm used in the setting of expander removal and implant positioning after mastectomy + RT
  Interventions: Device: acellular dermal matrix implant for breast reconstruction
- POST EXPANDER VERITAS: Veritas adm used in the setting of expander removal and implant positioning after mastectomy + RT
  Interventions: Device: acellular dermal matrix implant for breast reconstruction
- IMPLANT EXCHANGE NATIVE: Native adm used in the setting of implant exchange after mastectomy + RT
  Interventions: Device: acellular dermal matrix implant for breast reconstruction
- IMPLANT EXCHANGE VERITAS: Veritas adm used in the setting of implant exchange after mastectomy + RT
  Interventions: Device: acellular dermal matrix implant for breast reconstruction
- IMPANT EXCHANGE AFTER QUART NATIVE: Native adm used in the setting of implant exchange after QUART+ Mastectomy and implant reconstruction
  Interventions: Device: acellular dermal matrix implant for breast reconstruction
- IMPLANT EXCHANGE AFTER QUART VERITAS: Veritas adm used in the setting of implant exchange after QUART+ Mastectomy and implant reconstruction
  Interventions: Device: acellular dermal matrix implant for breast reconstruction

INTERVENTIONS:
Device: acellular dermal matrix implant for breast reconstruction — acellular dermal matrix implant in implant-based breast reconstruction in patients receiving radiotherapy

SUMMARY:
The goal of this retrospective observational trial is to compare two different devices, used in implant-based breast reconstruction, called acellular dermal matrices, which are a sort of collagen patch that integrates with the tissues of the patient and helps in contrasting the collateral effects of radiotherapy (capsular contracture, implant loss)

The main questions the study aims to answer are:

* is one of the two matrices better than the other? (better results with fewer complications)
* is there a group of patients who benefit more than another from the use of this type of devices?
* is there an adm which works better in one specific subgroup of patients? Participants have undergone mastectomy, radiotherapy and implant reconstruction with the aid of two different kinds of acellular dermal matrices.

Researchers will compare patients who receive the porcine-derived adm and the patients who receive bovine-derived adm to see if there is a difference in terms of capsular contracture reduction, aestethic result and complications.

DETAILED DESCRIPTION:
Radiotherapy is highly effective in breast cancer treatment, yet it impairs satisfactory implant-based reconstruction, due to high rates of capsular contracture and implant loss. This said, a fervent investigtion exists upon solutions that can make implant-based reconstruction safer and aesthetically satisfying, including the use of acellular dermal matrices. We retrospectively want to analyze our ADM-assisted post-RT implant-based breast reconstructions comparing two different matrices (porcine and bovine), when autologous reconstruction was contraindicated, to assess eventual differences in efficacy and risk profile of the devices. We want to further stratify the population in 4 groups based on clinical presentation to assess if there was a group where ADMs proves to perform better (Group A - previous quadrantectomy, Group B - previous mastectomy and expander reconstruction, Group C - previous mastectomy and implant reconstruction, Group D - prior quadrantectomy followed by mastectomy and implant reconstruction).

ELIGIBILITY:
Inclusion Criteria:

* at least 6 months follow up
* breast reconstruction with implant + acellular dermal matrix after mastectomy and radiotherapy

Exclusion Criteria:

* mastectomy flap <1 cm
* autoimmune disease
* prolonged use of corticosteroids

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — female patients undergoing breast reconstruction after mastectomy
Study Population: The study focuses on female patients undergoing implant based reconstruction after radiotherapy assisted by the use of an acellular dermal matrix.
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-10-13 (Actual)

PRIMARY OUTCOMES:
ADM efficacy and risk profile comparison | 60 months
  Does one dermal matrix perform better than the other in terms of efficacy and complication rates?

SECONDARY OUTCOMES:
Best clinical setting for ADM use | 60 months
  Is there a subgroup of patient where the use of ADM proves more beneficial than others?

OTHER OUTCOMES:
ADM comparison in each clinical setting group | 60 months
  Is there a type of dermal matrix that performs better than the other in a specific subgroup of patients?

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Vittorio Emanuele Lisa, MD, Principal Investigator — Istituto Europeo di Oncologia
Locations (1):
- European Institute of Oncology, Milan, Lombardy, Italy